CLINICAL TRIAL: NCT04117672
Title: Evaluation of Antisecretory Factor in Treatment of Severe Traumatic Brain Injury With Multimodal Monitoring
Brief Title: Antisecretory Factor In Severe Traumatic Brain Injury
Acronym: AFISTBI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter Siesjö (Other)
Collaborators: Skane University Hospital (Other); Lantmannen Medical AB (Other)
Responsible Party: Sponsor-Investigator, Peter Siesjö, Professor, Skane University Hospital
Organization: Skane University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-00553
Record Dates: First submitted 2019-09-23; First posted 2019-10-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; cerebral edema; antisecretory factor; inflammatory cytokines; cerebral oxygen monitoring; intracranial pressure; microdialysis
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Edema | interventions — antisecretory factor

STUDY DESIGN:
Intervention Model Description: Participants with severe TBI and scheduled for multimodal monitoring will be randomised to active or placebo treatment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Egg powder enriched for antisecretory factor and placebo egg powder with the same color, taste and texture,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Egg yolk powder not enriched for antisecretory powder
  Interventions: Dietary Supplement: Placebo egg yolk powder
- Salovum (Experimental): Egg yolk powder enriched for antisecretory powder
  Interventions: Dietary Supplement: Salovum

INTERVENTIONS:
Dietary Supplement: Salovum — Active egg yolk powder
  Other Names: Antisecretory factor
  Arms: Salovum
Dietary Supplement: Placebo egg yolk powder — Normal egg yolk powder
  Arms: Placebo

SUMMARY:
This study evaluates the addition of Salovum, an egg yolk powder enriched for antisecretory factor, to standard care of participants with severe traumatic brain injury. Half of the participants will be administered Salovum while the other half will be given a placebo egg yolk powder, not enriched for antisecretory factor. Intracranial pressure (ICP), partial brain oxygen pressure (PtbO2), microdialysis of metabolites and inflammatory mediators and trauma intensity level (TIL) will be assessed in all patients.

DETAILED DESCRIPTION:
Cerebral edema accounts for an essential part of the morbidity and mortality in severe traumatic brain injury but can also arise in other cerebral pathologies such as infectious and ischemic conditions such e.g. stroke and meningitis. Cerebral edema can lead to an elevated intracranial pressure (ICP) with impact on both perfusion and diffusion in the brain.

AF (antisecretory factor) is a 41 kilodalton endogenous and essential protein with proposed antisecretory and anti-inflammatory effects. AF is homologous to S5A and Rpn10 proteins which are parts of the 26S proteasome subunit. AF also shows close homology to angiocidin a protein with reported anti-proliferative and anti-angiogenic properties. The AF protein is cleaved into several active peptides, one of which has been synthesized within a 16 amino acid peptide (AF-16) that has been used in animal experimental studies. Salovum® is a product based on the egg yolk powder B221®, and contains high levels of AF. Salovum® is classified as a food for special medical purposes (FSMP) by the European Food Safety Agency.

AF has shown clinical effects in Mb Ménière, mastitis and meningitis. Experimentally AF-16 and AF have been shown to reduce intracranial pressure and improve outcome in models of traumatic brain injury (TBI) and herpes encephalitis. Preliminary results show reduction of ICP and improved outcome in human traumatic brain injury. A randomized, prospective, double-blinded phase 2-3 in participants with severe traumatic head injury is ongoing at Tygerberg University Hospital, Cape Town, South Africa (ClinicalTrials.gov identification number: NCT03339505).

The antisecretory factor is an endogenous protein and no antibody formation has been demonstrated in human administration. Although Salovum® has been given to hundreds of patients, no side effects have been recorded. Egg yolk allergy is a contraindication but no cases of triggered allergy have been reported.

The mechanisms underlying the effects of antisecretory factor on cerebral edema are not clarified. Immune modulation through effects on myeloid cells, proteasome modulation and effects on ion pumps have been proposed.

The present study intends to clarify mechanisms behind the proposed effect of antisecretory factor in cerebral edema In the present study participants with severe traumatic brain injury as defined in inclusion and exclusion criteria will be randomised to either treatment with Salovum or placebo egg powder during 5 days after enrolment. Randomisation will be performed in blocks and randomisation envelopes will be used with the number inside the envelope. Salovum and normal egg powder will be suspended with tap water and administered through the gastric feeding tube. All participants will receive standard care for severe TBI according to the treatment algorithm at the Neuro Intensive Care Unit (NICU), Department of Neurosurgery, Skåne University Hospital, Lund, Sweden. The algorithm prescribes invasive monitoring of ICP, PtbO2 and metabolites (cerebral microdialysis). As this algorithm includes stepwise co-interventions in order to control ICP and cerebral perfusion pressure (CPP) the TIL score will be used to compensate for the bias of increased co-interventions in either arm. At follow up patients will be assessed for mortality and Glasgow Outcome Scale-Extended (GOSE)

ELIGIBILITY:
Inclusion Criteria:

Severe traumatic brain injury, Glasgow Outcome Scale (GCS) <9 at admission to NICU.

Clinical indication for insertion of intracranial pressure monitor, intracerebral oxygen pressure monitor and microdialysis catheter.

Consultation with relatives or consent from guardians.

Exclusion Criteria:

Known egg yolk allergy.

Unilateral or bilateral fixed and dilated pupil after initial operative intervention.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
ICP mean | During intervention, 5 days
  Measured by an intracranial pressure sensor

SECONDARY OUTCOMES:
Concentration of inflammatory cytokines | During intervention, 5 days
  Interleukin-6 (Il-6), interleukin-8 (IL-8) and monocyte chemotactic protein (MCP-1) assessed from microdialysate and plasma by multiplex analysis

OTHER OUTCOMES:
Mortality | At 30 days and 12 months
  Mortality due to traumatic brain injury
Morbidity | At 6 and 12 months
  Assessed by Glagow Outcome Scale-Extended (GOSE). Minimum 1 (full recovery). MAXIMUM 8 (DEAD)
Intracerebral oxygen partial pressure | During intervention, 5 days
  Measured by an intracranial oxygen sensor
Intracerebral oxygen partial pressure | Change from baseline during intervention, up to 6 days
  Lactate/pyruvate ratio assessed by online microdialysis
Treatment intensity level | During intervention, 5 days
  Treatment intensity level (TIL) scale. Minimum 0 (no intervention to control intracranial pressure (ICP)), maximum 38 points (maximum efforts to control ICP)
Treatment intensity level | Change from baseline during intervention, up to 6 days
  Treatment intensity level (TIL) scale. Minimum 0 (no intervention to control intracranial pressure (ICP)), maximum 38 points (maximum efforts to control ICP)
Rate of cerebral metabolism | During intervention, 5 days
  Lactate/pyruvate ratio assessed by online microdialysis
Rate of cerebral metabolism | Change from baseline during intervention, up to 6 days
  Lactate/pyruvate ratio assessed by online microdialysis
Concentration of brain damage markers | During intervention, 5 days
  Glial fibrillary acidic protein (GFAP) and neuron-specific enolase (NSE) assessed from microdialysate and plasma
Concentration of brain damage markers | Change from baseline during intervention, up to 6 days
  Glial fibrillary acidic protein (GFAP) and neuron-specific enolase (NSE) assessed from microdialysate and plasma
ICP area under curve | During intervention, 5 days
  Measured by an intracranial pressure sensor
ICP area under curve | Change from baseline during intervention, up to 6 days
  Measured by an intracranial pressure sensor
ICP mean | Change from baseline during intervention, up to 6 days
  Measured by an intracranial pressure sensor
Concentration of inflammatory cytokines | Change from baseline during intervention, up to 6 days
  Interleukin-6 (Il-6), interleukin-8 (IL-8) and monocyte chemotactic protein (MCP-1) assessed from microdialysate and plasma by multiplex analysis

CONTACTS AND LOCATIONS:
Overall Officials: Peter Siesjö, MD, PhD, Principal Investigator — Skane University Hospital
Locations (1):
- Skane University Hopsital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data that underlie published results will be made available after publication.after de identification.
Supporting Information: Study Protocol
Time Frame: From 3 months after publication to 24 months after publication.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Background] Ilkhanizadeh S, Sabelstrom H, Miroshnikova YA, Frantz A, Zhu W, Idilli A, Lakins JN, Schmidt C, Quigley DA, Fenster T, Yuan E, Trzeciak JR, Saxena S, Lindberg OR, Mouw JK, Burdick JA, Magnitsky S, Berger MS, Phillips JJ, Arosio D, Sun D, Weaver VM, Weiss WA, Persson AI. Antisecretory Factor-Mediated Inhibition of Cell Volume Dynamics Produces Antitumor Activity in Glioblastoma. Mol Cancer Res. 2018 May;16(5):777-790. doi: 10.1158/1541-7786.MCR-17-0413. Epub 2018 Feb 5. PMID 29431617
- [Background] Clausen F, Hansson HA, Raud J, Marklund N. Intranasal Administration of the Antisecretory Peptide AF-16 Reduces Edema and Improves Cognitive Function Following Diffuse Traumatic Brain Injury in the Rat. Front Neurol. 2017 Feb 14;8:39. doi: 10.3389/fneur.2017.00039. eCollection 2017. PMID 28261150
- [Background] Lonnroth I, Oshalim M, Lange S, Johansson E. Interaction of Proteasomes and Complement C3, Assay of Antisecretory Factor in Blood. J Immunoassay Immunochem. 2016;37(1):43-54. doi: 10.1080/15321819.2015.1042544. PMID 25897558
- [Background] Al-Olama M, Lange S, Lonnroth I, Gatzinsky K, Jennische E. Uptake of the antisecretory factor peptide AF-16 in rat blood and cerebrospinal fluid and effects on elevated intracranial pressure. Acta Neurochir (Wien). 2015 Jan;157(1):129-37. doi: 10.1007/s00701-014-2221-7. Epub 2014 Sep 24. PMID 25248325
- [Background] Johansson E, Al-Olama M, Hansson HA, Lange S, Jennische E. Diet-induced antisecretory factor prevents intracranial hypertension in a dosage-dependent manner. Br J Nutr. 2013 Jun 28;109(12):2247-52. doi: 10.1017/S0007114512004552. Epub 2012 Nov 16. PMID 23153478
- [Background] Hansson HA, Al-Olama M, Jennische E, Gatzinsky K, Lange S. The peptide AF-16 and the AF protein counteract intracranial hypertension. Acta Neurochir Suppl. 2012;114:377-82. doi: 10.1007/978-3-7091-0956-4_73. PMID 22327727
- [Background] Jennische E, Bergstrom T, Johansson M, Nystrom K, Tarkowski A, Hansson HA, Lange S. The peptide AF-16 abolishes sickness and death at experimental encephalitis by reducing increase of intracranial pressure. Brain Res. 2008 Aug 28;1227:189-97. doi: 10.1016/j.brainres.2008.05.083. Epub 2008 Jun 11. PMID 18586012
- [Background] Lange S, Lonnroth I. The antisecretory factor: synthesis, anatomical and cellular distribution, and biological action in experimental and clinical studies. Int Rev Cytol. 2001;210:39-75. doi: 10.1016/s0074-7696(01)10003-3. PMID 11580208
- [Background] Johansson E, Lonnroth I, Lange S, Jonson I, Jennische E, Lonnroth C. Molecular cloning and expression of a pituitary gland protein modulating intestinal fluid secretion. J Biol Chem. 1995 Sep 1;270(35):20615-20. doi: 10.1074/jbc.270.35.20615. PMID 7657640
- [Derived] Reen L, Cederberg D, Marklund N, Visse E, Siesjo P. Antisecretory factor in severe traumatic brain injury (AFISTBI): protocol for an exploratory randomized placebo-controlled trial. Trials. 2025 Feb 7;26(1):43. doi: 10.1186/s13063-025-08760-7. PMID 39920739